CLINICAL TRIAL: NCT01436448
Title: Effects of Probiotics (Lactobacillus Rhamnosus) In Reducing Glucose Intolerance During and After Pregnancy: A Double Blind Randomized Controlled Trial in Antenatal Clinic of Karachi-Pakistan (GRIP)
Brief Title: Probiotics (Lactobacillus Rhamnosus) in Reducing Glucose Intolerance During and After Pregnancy
Acronym: GRIP
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Aga Khan University (Other)
Responsible Party: Principal Investigator, Bilal Ahmed, Senior Instructor Research, Aga Khan University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 111012MED
Record Dates: First submitted 2011-09-07; First posted 2011-09-19 (Estimated); Last update posted 2011-09-20 (Estimated); Status verified 2011-09

CONDITIONS: Glucose Intolerance; Pregnancy
Keywords: efficacy; Lactobacillus Rhamnosus; glucose intolerance; feasibility; compliance and safety; reducing glucose intolerance during and after pregnancy
MeSH Terms: conditions — Glucose Intolerance; Patient Compliance

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Probiotics Lactobacillus Rhamnosus (Experimental): dose of 1010 Colony forming Units (CFU) once daily till delivery will be given orally
  Interventions: Drug: Probiotics Lactobacillus Rhamnosus
- Placebo (No Intervention): Microcrystalline cellulose/d each, up till deliver

INTERVENTIONS:
Drug: Probiotics Lactobacillus Rhamnosus — Probiotics Lactobacillus Rhamnosus (1010 Colony forming Units (CFU)/day)
  Arms: Probiotics Lactobacillus Rhamnosus

SUMMARY:
Introduction: The overall aim of the study is to assess the efficacy of Lactobacillus Rhamnosus in reducing glucose intolerance during and after pregnancy. A second objective of the study is to determine the feasibility, compliance and safety of Lactobacillus Rhamnosus among this cohort. Within this goal is to determine whether the investigators can enroll women at high risk for developing Gestational Diabetes Mellitus (GDM) and follow them out at regular antenatal visits and 6-weeks post partum.

Women with GDM are, 7 times more at risk of developing type 2 diabetes compared with those who had a normo- glycaemic pregnancy. The population attributable risk for type 2 diabetes mellitus (DM) in women with GDM is high, and around 30 - 50% women with GDM converts into type 2 (DM) which is associated with pre-mature morbidity, mortality and high economic burden. It is evident that untreated GDM is associated with higher incidence of complications during pregnancy and increases the risk of perinatal mortality and infant morbidity. The prevalence of GDM in Pakistan is around 8%, comparatively higher than other South Asian countries. Therefore, interventions that can improve glucose regulation during pregnancy are highly important.

Probiotics, the live micro-organisms, have shown promising results in regulating glucose metabolism among pregnant mice. The effect of Probiotics on glucose metabolism is attributable to their immuno-regulatory properties. They elicit powerful anti-inflammatory capabilities by inhibiting the NF-kB pathway, which mediates microbial activation of the immune system. Further, they diminish both fermentation of polysaccharides and induction of fasting-induced adipocyte factor gene transcription. The safety of Lactobacillus Rhamnosus among pregnant women is already established in other diseases.

A placebo controlled trial from Finland on pregnant females randomized to receive either dietary counseling and Probiotics (Lactobacillus Rhamnosus), concluded improved glucose tolerance as compared to the placebo group [OR 0.31 (95% CI 0.12, 0.78)]. However, this study could not determine the sole effects of probiotics in reducing glucose intolerance. Nevertheless, no studies on the role of Lactobacillus Rhamnosus in regulating glucose intolerance have been conducted in any other part of the world yet. Therefore, a pilot trial to see the efficacy, compliance and feasibility of Lactobacillus Rhamnosus among pregnant females is imperative. The objectives of the investigators study are:

* To assess the efficacy of Probiotics Lactobacillus Rhamnosus (1010 Colony forming Units (CFU)/day) in reducing glucose intolerance among pregnant women attending antenatal clinic of Karachi-Pakistan.
* To assess the feasibility, compliance and safety of conducting a double blind, placebo controlled randomized trial of Lactobacillus Rhamnosus by recruiting high risk women during pregnancy attending antenatal clinics and following them up 6 weeks postpartum in Karachi-Pakistan.

Methods: For the pilot trial, women will be recruited from antenatal hospital of the city, during 12-14 weeks of gestation.

Study Design: The study will be double blind randomized, placebo controlled trial. Randomization will be done by blocked method. The dose of 1010 Colony forming Units (CFU) once daily till delivery will be given orally.

Study Endpoints and Ascertainment: Baseline information will be comprised of socioeconomic status, parity, gravida, blood pressure and obstetric history etc. The study endpoint comprises of efficacy, feasibility, compliance and safety and will be ascertained at monthly follow-up, during week 24 - 28, and 6 weeks post partum. Efficacy will be ascertained by Oral Glucose Tolerance Test (OGTT) performed at randomization and during 24-28 weeks of gestation. Feasibility and compliance will be assessed through recruitment rate, drop-out rate, reasons for drop-out, non-participation and empty drug sachet count.

ELIGIBILITY:
Inclusion Criteria:

High risk pregnancy ( presence of more than or equal to 1 of the following)

* Maternal age greater than or equal to 35
* Family history of diabetes among 1st degree relative defined as parents, siblings and children
* Overweight (BMI greater than 23) Women visiting the antenatal clinics during 12-14 weeks of gestation Women with Singleton pregnancy Women whose delivery is planned at the study hospital

Exclusion Criteria:

* History of GDM ( since in our setting the women are not usually screen for pre- gestational diabetes therefore it is difficult to differentiate between GDM and pre gestational diabetes)
* Known Diabetes mellitus
* Known chronic diseases ( hypothyroidism ,cardiac, renal, rheumatoid arthritis, carcinoma)
* Women maintained on medications such as: corticosteroids, Azathioprin, antiepileptic epileptic drugs.
* Known Poly Cystic Ovarian Syndrome
* Non-residents of Karachi

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2011-10; Primary Completion 2012-11 (Estimated); Study Completion 2013-05 (Estimated)

PRIMARY OUTCOMES:
Glucose Intolerance | 24-28 weeks of pregnancy
  Glucose Intolerance. Glucose intolerance will be assessed in accordance with ADA guidelines by OGTT. OGTT will be performed during 24-28 weeks of pregnancy
Glucose Intolerance | 6 to 8 weeks post partum
  Glucose Intolerance. Glucose intolerance will be assessed in accordance with ADA guidelines by OGTT. OGTT will be performed during 6 to 8 weeks post partum

SECONDARY OUTCOMES:
Feasibility | 36 weeks
  * Process of recruitment rate assessed at monthly antenatal visit
  * recruitment rate rate assessed at monthly antenatal visit
  * Reasons for non-participation rate assessed at monthly antenatal visit
Compliance | 36 weeks
  * the compliance rate assessed at monthly antenatal visit
  * side effects rate assessed at monthly antenatal visit
  * drop-out rate rate assessed at monthly antenatal visit
  * reasons for drop-out rate assessed at monthly antenatal visit
Maternal safety | at the time of delivery till 42 weeks postpartum
  MATERNAL OUTCOMES:( :( assessed at the time of delivery and postpartum)
  Maternal Mortality Maternal Weight Gain Preeclampsia Induction of labor Mode of Delivery
FETAL/NEONATAL safety | assessed at the time of delivery till 6-8 weeks postpartum
  Death This will include:
  Still births Neonatal death Pre-term birth. Birth Trauma Macrosomia Small for Gestational Age Polyhydramnios Recurrent Hypoglycemia Large for Gestational Age Shoulder Dystocia 5-minute Apgar score: <7 Hyperbilrubinemia Respiratory Distress NICU Admission

CONTACTS AND LOCATIONS:
Overall Officials: Bilal Ahmed, MSc, Principal Investigator — Aga Khan University; Abdul Jabbar, MBBS, FRCP, Study Chair — Aga Khan University; Kashmira Nanji, MSc, Principal Investigator — Aga Khan University; Ali Khowaja, FRCS — Aga Khan University; Sarah Saleem, MBBS, MSc — Aga Khan University; Rozina Sikandar, MBBS, FCPS — Aga Khan University
Locations (1):
- Aga Khan Hospital for Garden, Karachi, Sindh, Pakistan

REFERENCES:
- [Derived] Davidson SJ, Barrett HL, Price SA, Callaway LK, Dekker Nitert M. Probiotics for preventing gestational diabetes. Cochrane Database Syst Rev. 2021 Apr 19;4(4):CD009951. doi: 10.1002/14651858.CD009951.pub3. PMID 33870484